CLINICAL TRIAL: NCT04702516
Title: The Effect of Semaglutide (Ozempic) on Bone Turnover in Patients With Increased Fracture Risk: a Randomized Placebo-controlled Clinical Trial
Brief Title: The Effect of Semaglutide on Bone Turnover in Patients With Increased Risk of Bone Fracture
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Frost (Other)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Morten Frost, Associate professor, clinical staff specialist, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-20200048; 2020-000616-29 (EudraCT Number); 0052699 (Other Grant/Funding Number: Novo Nordisk Foundation); 18/51856 (Other Grant/Funding Number: Region of Southern Denmark); A35844 (Other Grant/Funding Number: Gangsted Foundation)
Record Dates: First submitted 2020-12-09; First posted 2021-01-11 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Ozempic 1 mg (or highest tolerated dose) s.c. once weekly for 52 weeks (incl. titration)
  Interventions: Drug: Ozempic
- Placebo (Placebo Comparator): Placebo (saline) 1 mg (or highest tolerated dose) s.c. once weekly for 52 weeks (incl. titration)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozempic — 2 mg prefilled pen for subcutaneous injection, 0.25 mg for two weeks then 0.5 mg for two weeks and then 1 mg for another 48 weeks.
  Arms: Semaglutide
Drug: Placebo — 2 mg prefilled pen for subcutaneous injection, 0.25 mg for two weeks then 0.5 mg for two weeks and then 1 mg for another 48 weeks.
  Arms: Placebo

SUMMARY:
The hypothesis for this study is that the GLP-1Ra Semaglutide has a positive effect on the balance between build-up and degradation as well as the strength of the bones in men and women aged 40-85 years at increased risk of bone fractures. Treatment involves injection of Semaglutide 1.34 mg/ml once a week or corresponding volume of placebo once a week for 52 weeks. The effect will be measured by bone markers in blood samples, bone scans, bone tissue tests (bone biopsy), and direct bone strength measured by microindentation at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* T-score <-1 in hip or lower back, assessed by DXA scan and / or
* Low-energy fracture within the last 3 years

Exclusion Criteria:

* T-score <-2.5 in hip or lower back, assessed by DXA scan, although these individuals may be included if they prefer to participate or are not candidates for conventional therapy, e.g., by eGFR <35 or adverse reaction (influenza-like symptoms, allergic reaction, etc.) to, e.g., bisphosphonate therapy
* Diabetes type 1 and 2
* Heart failure similar to NYHA Class IV
* Primary hyperparathyroidism
* Vitamin D deficiency (<25 nM) (re-test after substitution acceptable)
* Known disorders affecting bone metabolism, e.g., uncontrolled thyrotoxicosis, severe renal impairment (eGFR <20) or liver function (baseline phosphatase higher than twice upper limit (105 U/L)), rheumatism, celiac disease, hypogonadism, severe COPD, hypopituitarism, Cushing's disease
* Antiresorptive or bone anabolic drugs for the last 12 months
* Use of anabolic steroids in the previous year
* History of pancreatitis
* Allergy to the medicines used
* Inability to give informed consent
* BMI <20 kg / m2

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Procollagen type 1 N-terminal propeptide (P1NP) | Baseline and 52 weeks
  Percentage changes in bone formation marker P1NP from baseline and after 12 months

SECONDARY OUTCOMES:
Collagen 1 cross link C-terminal telopeptide (CTX) | Baseline and 52 weeks
  Changes in bone resorption marker CTX from baseline and after 12 months
Tartrate-resistant acid phosphatase (TRAP) | Baseline and 52 weeks
  Changes in bone resorption marker TRAP from baseline and after 12 months
Osteocalcin | Baseline and 52 weeks
  Changes in bone formation marker osteocalcin from baseline and after 12 months
Bone specific alkaline phosphatase (BALP) | Baseline and 52 weeks
  Changes in bone formation marker BALP from baseline and after 12 months
BMSi | Baseline and 52 weeks
  Changes in direct bone strength measured by microindentation from baseline and after 12 months
Bone mineral density (BMD) | Baseline and 52 weeks
  Changes in BMD (total hip, femoral neck and lumbar spine (L1-4)) assessed by DXA scans from baseline and after 12 months
Estimated bone strength | Baseline and 52 weeks
  Changes in estimated bone strength assessed by finite elemental analysis (HR-pQCT scan) from baseline and after 12 months
Total volumetric BMD | Baseline and 52 weeks
  Changes in total volumetric BMD (mg/cm^3) assessed by HR-pQCT scan of distal tibia and radius
Trabecular volumetric BMD | Baseline and 52 weeks
  Changes in trabecular volumetric BMD (mg/cm^3) assessed by HR-pQCT scan of distal tibia and radius
Cortical volumetric BMD | Baseline and 52 weeks
  Changes in cortical volumetric BMD (mg/cm^3) assessed by HR-pQCT scan of distal tibia and radius
Bone volume | Baseline and 52 weeks
  Changes in trabecular bone volume pr total volume (BV/TV) assessed by HR-pQCT scan of distal tibia and radius
Trabecular thickness | Baseline and 52 weeks
  Changes in trabecular thickness (mm) assessed by HR-pQCT scan of distal tibia and radius
Cortical thickness | Baseline and 52 weeks
  Changes in cortical thickness (mm) assessed by HR-pQCT scan of distal tibia and radius
Cortical porosity | Baseline and 52 weeks
  Changes in cortical porosity assessed by HR-pQCT scan of tibia and radius
Bone formation rate | 52 weeks
  Changes in bone formation rate (BRF/BS, µm^3/µm^2 per day), the volume of mineralized bone made per unit surface of bone per year

OTHER OUTCOMES:
Mirco RNAs | Baseline and 52 weeks
  Changes in expression of blood-circulating microRNAs (miRNAs) known to be involved in regulation of bone formation and bone resorption using qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Morten Frost, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Derived] Hansen MS, Wolfel EM, Jeromdesella S, Moller JK, Ejersted C, Jorgensen NR, Eastell R, Hansen SG, Frost M. Once-weekly semaglutide versus placebo in adults with increased fracture risk: a randomised, double-blinded, two-centre, phase 2 trial. EClinicalMedicine. 2024 May 3;72:102624. doi: 10.1016/j.eclinm.2024.102624. eCollection 2024 Jun. PMID 38737002